CLINICAL TRIAL: NCT04588571
Title: Efficacy and Safety Comparison of the Open (Femoral-popliteal Proximal Bypass) and Endovascular (Recanalization With Angioplasty and Stenting With Biomimetic Interwoven Nitinol Stent) Surgical Methods for the Treatment of Long Atherosclerotic Lesions of the Femoral-popliteal Segment Above the Knee, TASC II, Type D
Brief Title: Efficacy and Safety Comparison of the Open Surgical and Endovascular Methods for the Treatment of Long Atherosclerotic Lesions of the Femoral-popliteal Segment Above the Knee, TASC II, Type D.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sosudi2
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Atherosclerosis; Ischemia Limb; Superficial Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: interwoven nitinol stent; atherosclerosis; prolonged occlusion of SFA; endovascular treatment; femoro-popliteal bypass; TASC II, type D
MeSH Terms: conditions — Atherosclerosis | interventions — Angioplasty; Stents

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, open-label study. Group 1 (n=55): Femoropopliteal proximal bypass. Group 2 (n=55): Recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular treatment (Experimental): Patients (n=55) with recanalization of the femoral-popliteal arterial segment (TASC II, type D) above the knee with a biomimetic braided nitinol stent.
  Interventions: Procedure: Endovascular recanalization with angioplasty and stenting with the biomimetic interwoven nitinol stent
- Open surgery (Active Comparator): Patients (n=55) with femoropopliteal proximal bypass with a prolonged atherosclerotic lesion of the femoropopliteal arterial segment (TASC II, type D).
  Interventions: Procedure: Femoropopliteal proximal bypass

INTERVENTIONS:
Procedure: Endovascular recanalization with angioplasty and stenting with the biomimetic interwoven nitinol stent — Under local anesthesia, a standard endovascular approach is performed and the affected arterial segment is visualized. Transluminal or subintimal recanalization of the occluded arterial segment is performed with a hydrophilic guidewire. Next, balloon angioplasty of the recanalized segment is performed. After control angiography, a biomimetic interwoven nitinol stent is placed throughout the lesion.
  Drug therapy includes pre-procedure aspirin (160-300 mg/day), starting at least one day before, and intra-procedure heparin (100 U / kg body weight intravenously). After the procedure, all patients have prescribed aspirin (100 mg per day) for a long time and clopidogrel (75 mg per day) for 3 months.
  Arms: Endovascular treatment
Procedure: Femoropopliteal proximal bypass — Under general anesthesia, 2 standard open surgical approaches are performed: first - to the common femoral artery, superficial femoral artery, and deep femoral artery; the second - to the first portion of the popliteal artery. After systemic heparinization, clamps are applied to the arteries. A longitudinal arteriotomy of the popliteal artery is performed, and a distal end-to-side anastomosis is formed between the artery and the shunt. Next, the shunt is passed into the groin wound. Longitudinal arteriotomy of the common femoral artery. A proximal end-to-side anastomosis is formed between the shunt and the common femoral artery. Surgical hemostasis wound drainage and layer-by-layer wound closure are performed.
  Drug therapy includes pre-procedure aspirin (160-300 mg/day), starting at least one day before, and intra-procedure heparin (100 U / kg body weight intravenously). After the procedure, all patients have prescribed aspirin (75-100 mg per day) for a long time.
  Arms: Open surgery

SUMMARY:
Endovascular revascularization and open bypass grafting above the knee show comparable results in primary 2-year patency (about 65%) in medium-length lesions - TASC II, C (Pereira et al, 2006). At the same time, a recent study, where the authors studied the effectiveness of stenting of long lesions (200 mm or more) of the chronic occlusions of the femoropopliteal segments (TASC II, D), showed unsatisfactory results (primary patency 45%) of the stented segment within 2 years (Lin et al, 2015). One of the possible solutions to the problem of breakage of stents in the femoral-popliteal position is a modified method of their manufacture by braiding from nitinol wire. Some studies with intervowen nitinol stents did show their resistance to breakage in this position. Moreover, the primary patency was > 70%. (Werner et al, 2014). These data suggest a better primary patency rate within 2 years with a longer lesion length (>200 mm).

This is a prospective, randomized, open-label study. The main objective of the study is to compare the clinical efficacy and safety of two therapies for the treatment of prolonged atherosclerotic lesions of the arteries of the femoropopliteal segment above the knee, TASC II type D - femoropopliteal proximal shunting and recanalization with angioplasty and stenting using biomimetic interwoven nitinol stent in patients with symptomatic peripheral arterial disease at 24 months. Secondary objectives are to identify predictors of restenosis and occlusions of the operating segment and compare the quality of life of patients after the procedure. It is planned to recruit 110 patients (55 patients in each group). Observation period 2 years. Primary endpoint:

-The effectiveness of the method of surgical treatment after 24 months (primary patency, primary-assisted patency, secondary patency).

Secondary endpoints:

* Clinical efficacy of the method of surgical treatment after 24 months (MALE);
* Safety of the method of surgical treatment in the early postoperative period (hematoma of the surgical access area, peripheral neuropathy, purulent-infectious complications of the surgical access area) and after 24 months (MACE);
* Assessment of the quality of life in patients after surgical treatment at 6, 12, and 24 months (SF-36 questionnaire);
* Evaluation of prognostic factors for adverse outcomes after surgical treatment.

DETAILED DESCRIPTION:
Endovascular revascularization and open bypass grafting above the knee show comparable results in primary 2-year patency (about 65%) in medium-length lesions - TASC II, C (Pereira et al, 2006). At the same time, a recent study, where the authors studied the effectiveness of stenting of long lesions (200 mm or more) of the chronic occlusions of the femoropopliteal segments (TASC II, D), showed unsatisfactory results (primary patency 45%) of the stented segment within 2 years (Lin et al, 2015). One of the possible solutions to the problem of breakage of stents in the femoral-popliteal position is a modified method of their manufacture by braiding from nitinol wire. Some studies with interwoven nitinol stents did show their resistance to breakage in this position. Moreover, the primary patency was > 70%. (Werner et al, 2014). These data suggest a better primary patency rate within 2 years with a longer lesion length (>200 mm).

This is a prospective, randomized, open-label study. The main objective of the study is to compare the clinical efficacy and safety of two therapies for the treatment of prolonged atherosclerotic lesions of the arteries of the femoropopliteal segment above the knee, TASC II type D - femoropopliteal proximal shunting and recanalization with angioplasty and stenting using biomimetic interwoven nitinol stent in patients with symptomatic peripheral arterial disease at 24 months. Secondary objectives are to identify predictors of restenosis and occlusions of the operating segment and compare the quality of life of patients after the procedure.

The analysis of literature data showed, that two-year primary patency after endovascular revascularization using a nitinol stent in long lesions was 60%. At the same time, the two-year primary patency after the femoropopliteal proximal bypass was 56% (Enzmann et al. Nitinol stent versus bypass in long femoropopliteal lesions: 2-year results of a randomized controlled trial. JACC: Cardiovascular Interventions. 2019 Dec 23; 12 (24): 2541-9.). Considering these data, it should be assumed that the use of biomimetic interwoven nitinol stents will slightly improve the primary patency parameters within 2 years in the stenting group. The 2-year primary patency after stenting of the femoropopliteal segment with an interwoven nitinol stent was 76% (Scheinert et al., 2011). A power analysis was performed to calculate the sample size of the "non-inferiority" design for a study power of 80%, a type 1 error probability of 5%, and a non-inferiority margin of 10%. It is planned to recruit 110 patients (55 patients in each group). The observation period of 2 years. Primary endpoint:

-The effectiveness of the method of surgical treatment after 24 months (primary patency, primary-assisted patency, secondary patency).

Secondary endpoints:

* Clinical efficacy of the method of surgical treatment after 24 months (MALE);
* Safety of the method of surgical treatment in the early postoperative period (hematoma of the surgical access area, peripheral neuropathy, purulent-infectious complications of the surgical access area) and after 24 months (MACE);
* Assessment of the quality of life in patients after surgical treatment at 6, 12, and 24 months (SF-36 questionnaire);
* Evaluation of prognostic factors for adverse outcomes after surgical treatment. Screening It is performed in patients with a verified diagnosed occlusive lesion of the femoropopliteal segment above the knee joint (type D according to the TASC II classification), with chronic ischemia of the lower extremities of 3-6 categories according to Rutherford.

  * Assessment of inclusion/exclusion criteria
  * Assigning a patient number

Study inclusion Collecting baseline information about the patient (history, including information about concomitant therapy, data from the initial physical examination, ultrasound data of the lower limb arteries, CT -arteriography data, assessment of the quality of life using the SF-36 questionnaire. Randomization using the envelope method to one group or another.

Group 1: Femoropopliteal proximal bypass; Group 2: Recanalization of prolonged occlusion of the arteries of the femoral-popliteal segment above the knee joint with angioplasty and stenting with a biomimetic interwoven nitinol stent.

Follow up period; 6, 12, and 24 months.

Performed:

Triplex ultrasound of one lower limb (restenosis, thrombosis, stent breakage);

* Leg's roentgenography for the stenting group in two projections, for patients in whom a stent breakage is suspected according to ultrasound;
* Consultation with a cardiovascular surgeon.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* Symptomatic lesion (Rutherford category 3 - 6);
* Atherosclerotic prolonged occlusive lesion of the femoropopliteal arterial segment above the knee, classified by TASC II as type D, confirmed by computed tomography or arteriography;
* De novo lesion;
* Patient informed consent.

Exclusion Criteria:

* Age < 18 years old;
* Potentially pregnant women;
* Asymptomatic lesion;
* Acute ischemia;
* Not de novo lesion;
* Severe comorbidity with a life expectancy of fewer than 2 years;
* Contraindications to antiplatelet therapy (double antiplatelet therapy is required for at least 2 months after the intervention);
* Patient participation in another clinical trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
primary patency | 24 months
  primary patency is defined as absence of occlusion or flow-limiting stenosis (peak systolic velocity [PSV] ratio >2.5) of the treated segment including 1 cm proximal and distal of the anastomosis.
primary assisted patency | 24 months
  primary assisted patency is defined as a secondary procedure is performed to prevent failure (in a flow-limiting stenosis [PSV ratio >2.5] in a still-patent segment of stent or bypass, including the anastomoses.
secondary patency | 24 months
  secondary patency is defined as a secondary procedure performed for graft or stent occlusion in an afterward patent vessel.

SECONDARY OUTCOMES:
MALE | 24 months
  Major adverce limb events
Safety of the surgical treatment in the early postoperative period | 30 days
  hematoma of the surgical access area, peripheral neuropathy, purulent-infectious complications of the surgical access area
MACE | 24 months
  major adverce cardiovascular events, deaths
Assessment of the quality of life | 24 months
  SF-36 questionary

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin Research Institute of Pathology of Circulation, Novosibirsk, Novosibirsk Area, Russia